CLINICAL TRIAL: NCT06124209
Title: Use of Fibrin Sealant Patch for Vein Anastomosis During Deceased Donor Liver Transplantation- Randomized Clinical Trial
Acronym: HemoCava
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Paweł Rykowski, MD, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BVI_202301
Record Dates: First submitted 2023-11-03; First posted 2023-11-09 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Liver Transplant; Complications
Keywords: tachosil; liver transplantation; vena cava inferior anastomosis; fibrin sealant; hemostasis
MeSH Terms: interventions — TachoSil

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tachosil® used in Vena Cava Inferior anastomosis (Experimental): Tachosil® used in Vena Cava Inferior anastomosis.
  Interventions: Drug: TachoSil
- Control (No Intervention): Standard haemostatic treatment in HPB surgery.

INTERVENTIONS:
Drug: TachoSil — TachoSil used in Vena Cava Inferior anastomosis during liver transplantation.
  Other Names: fibrin sealant matrix; EU/1/04/277/001; TachoSil 9,5 x 4,8 cm; Collagen-Fibrin Patch
  Arms: Tachosil® used in Vena Cava Inferior anastomosis

SUMMARY:
The study aims to evaluate the effect of the hemostatic matrix with fibrinogen and thrombin (TachoSil®) on vena cava inferior anastomoses during liver transplantation from a deceased donor.

The research comprises two groups: an experimental cohort with patients receiving a hemostatic matrix of fibrinogen and thrombin on the anastomotic line of the inferior vena cava, and a control cohort utilizing hemostasis without matrix sealent. The study involves a total of 170 participants, evenly distributed with 85 patients in each group.

DETAILED DESCRIPTION:
Studies have shown that materials containing fibrin shorten the time to hemostasis in the case of planned liver resection, but did not show a significant effect on the occurrence of postoperative bleeding. The aim of the study is to supplement knowledge about hemostatic matrices in liver transplantation, which will be used for the inferior vena cava anastomosis.

The study aims to evaluate the effect of the hemostatic matrix with fibrinogen and thrombin (TachoSil®) on vena cava inferior anastomoses during liver transplantation from a deceased donor.

The research comprises two groups: an experimental cohort with patients receiving a hemostatic matrix of fibrinogen and thrombin on the anastomotic line of the inferior vena cava, and a control cohort utilizing hemostasis without matrix sealent. The study involves a total of 170 participants, evenly distributed with 85 patients in each group.

ELIGIBILITY:
Inclusion Criteria:

* age over 18
* elective liver transplantation
* informed consent to participate in the study

Exclusion Criteria:

-decision to use packing during liver transplantation (bail out strategy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2023-11-04 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Significant postoperative bleeding | 10 days
  occurrence of significant postoperative bleeding within 10 days after surgery, defined as the occurrence of one of the following:
  1. occurrence of hematoma larger than 100ml
  2. transfusion of packed red blood cells after surgery
  3. performing relaparotomy due to bleeding

SECONDARY OUTCOMES:
Postoperative complication | 10 days
  Occurance of complication assesed in Clavien-Dindo scale

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Rykowski, MD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Department of General Transplant and Liver Surgery, Warsaw, Mazovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
Anonimized IPD would be shared after personal contact, after PI approval
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: 5 years after study finish
Access Criteria: scintific puropse only